CLINICAL TRIAL: NCT06385613
Title: The Effect of Mobile-Based Education on Self-Care, Quality of Life and Complications in Patients With Intestinal Stoma
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Nilgun Soylemez, Lecturer, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: TDK-2024-13377
Record Dates: First submitted 2024-04-19; First posted 2024-04-26 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Intestinal Stoma Site Hemorrhage; Intestinal Stoma Leakage; Life Style, Healthy
Keywords: intestinal stoma; mobile-based education; self-care; quality of life; complication

STUDY DESIGN:
Intervention Model Description: Groups will be divided into control and intervention. People in the group will be randomly assigned in a simple randomized manner.
Who Masked: Participant
Masking Description: Individuals assigned to controls and interventions will not know which group they are in.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Experimental): Patients who have undergone stoma surgery will be divided into two groups as control and intervention by simple randomization. Patients assigned to the control group will receive standard stoma care training applied by the clinic. Patients will be met before surgery and necessary information will be obtained. A total of 5 interviews will be conducted with patients in both groups.
  Interventions: Behavioral: Mobile-based stoma care education group
- Mobile-based stoma care education group (Experimental): Patients who have undergone stoma surgery will be divided into two groups as control and intervention by simple randomization. Patients assigned to mobile-based stoma care education groupwill receive mobile-based stoma care training prepared by the researcher. Patients will be met before surgery and necessary information will be obtained. A total of 5 interviews will be conducted with patients in both groups.
  Interventions: Behavioral: Mobile-based stoma care education group

INTERVENTIONS:
Behavioral: Mobile-based stoma care education group — Individuals included in the intervention group will be given mobile-based stoma care trainings before surgery, on the 3rd postoperative day, on the day of discharge, and on the 1st and 3rd months after discharge, and their effectiveness will be measured using data collection forms.

SUMMARY:
Stomas are most commonly used in the gastrointestinal tract as ileostomy or colostomy. Although colorectal cancers are the most important factor causing intestinal stoma opening, intestinal ostomies are also used in cases such as congenital anomalies, obstructive or inflammatory bowel diseases, traumas requiring surgery, large defects caused by colorectal injuries as well as sigmoid colon volvulus and ischemic colitis. In stoma surgery performed to increase the duration and quality of life of individuals, the patient's compliance with the stoma and awareness of possible complications are important. Conditions such as peristomal skin problems, noisy bowel movements, stool leakage and pain make it difficult to adapt to the stoma.In addition, despite all the advances in stoma care products and surgical techniques, individuals are faced with stoma complications. Therefore, individuals with stoma should be closely monitored for complications. Inappropriately selected stoma site or bag/adapter system, lack of knowledge and skills related to stoma care can be listed among the possible causes of complications. Complications such as edema, bleeding, ischemia and mucocutaneous separation may develop in the first days after stoma surgery. In studies evaluating patients in terms of stoma compliance and complications in the literature, it has been observed that mobile-based trainings given to patients increase their stoma compliance and reduce the incidence of complications. With the mobile-based training planned to be used in the study, it is thought to contribute to the ability of individuals to perform stoma care independently. With the decrease in peristomal skin lesions and stoma complications, it is predicted that the quality of life of patients with stoma will increase, self-care competence will be formed, and health expenditures and therefore national health expenditures will decrease. It is thought that this mobile training application will not only provide support to patients with stoma but also guide healthcare professionals. It will also contribute to closing the shortage of stoma and wound care nurses in hospitals.

DETAILED DESCRIPTION:
There are many factors that make it difficult for individuals to adapt and cope with the stoma. The most important components in the prevention and treatment of complications can be listed as marking the stoma site, evaluation of the peristomal skin, placement and removal of the appropriate bag/adapter system with the correct technique, close monitoring of patients, patient education, and performing medical and surgical interventions. Nursing care; complication management, patient care, nutrition, excretion, family relations, sexuality, sexuality, worship, work life, social life should be carried out by determining the problems related to the areas and paying attention to the privacy areas. In this context, nursing care should include a care process that starts at the time of hospitalization and covers the post-discharge period. Nursing care should aim to diagnose problems, increase stoma compliance and quality of life, physical/psychological recovery and gain stoma care skills.

Easy access to online information presents a dichotomy in terms of risk and benefit. If the patient is unable to assess the quality of the information and its relevance for his/her specific situation, decision-making may be negatively affected, leading to negative outcomes. The benefit of digital communication, especially in the context of individuals with ostomies, is that it provides individuals, families and communities with scientific information about informed practices. This allows the individual to identify and indicate early signs of complications. They can also receive guidance on their problems, contributing to an easier and more appropriate decision-making process. Providing adequate stoma care enables patients to cope better with their stoma and is therefore important for improving their quality of life. Although the importance of stoma care has been reported, it remains inadequate in many aspects. Innovative mobile applications have a significant potential to overcome these shortcomings. self-efficacy and participation in care can be improved by using mobile applications. It has been stated that patients supported by mobile applications are better supported in stoma care and have more self-efficacy, so individuals receiving support will have a good quality of life.In a study conducted in Turkey, it was reported that individuals who used a mobile application had higher levels of stoma compliance, ability to care for the stoma on their own, and satisfaction with the training they received than those who used a printed booklet. However, it was stated that the application was not effective in preventing peristomal skin lesions. It was stated that additional studies are needed to determine which features of a mobile application may be useful in preventing such lesions. For this reason, it is thought that the mobile-based training application to be developed will contribute to the patients to accept and manage the process faster, to have competence in stoma care, and to perform stoma care independently with well-managed care and education.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand and speak Turkish,
* Not visually or hearing impaired,
* No neurological disease affecting psychiatric or cognitive status,
* Decision to perform ileostomy or colostomy,
* No previous experience with intestinal stoma,
* Patients who can use telephone and internet will be included in the study.

Exclusion Criteria:

* Don't lose your life
* Development of a serious complication after surgical intervention

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-06-22 (Estimated); Primary Completion 2025-04-22 (Estimated); Study Completion 2025-08-22 (Estimated)

PRIMARY OUTCOMES:
Adaptation of Quality Life Scale | Average 3 months after completion of stoma care education.
  Patients' quality of life with stoma will be evaluated.The scale consists of 21 items developed by Baxter et al. in 2006. The Turkish validity and reliability study of the scale was conducted by Karadağ, Öztürk and Çelik in 2011. The first two items of the scale score an individual's general satisfaction with his/her life between ''0'' and ''100'' (0 indicates complete dissatisfaction, 100 indicates complete satisfaction). The other items are grouped into three sub-dimensions. These dimensions are work/social life, sexuality/body image and stoma function, respectively. The scale also includes 1 item on economic status and 1 item on skin irritation, which are not included in any sub-dimension. Except for the first two items of the scale, the other 19 items are in the form of 5-point Likert scale as 1: never, 2: rarely, 3: occasionally, 4: often, and 5: always. Each sub-dimension is evaluated out of 100 points (0 indicates poor quality of life, 100 indicates good quality of life).
Ostomy Self-Care Index | Average 3 months after completion of stoma care education.
  The "Ostomy Self-Care Index" scale was developed by Giulia Villa et al. in 2019 to measure the self-care of patients with stoma. The Turkish validity and reliability of the scale was conducted by Avcu and Yıldız in 2022. The "Ostomy Self-Care Index" scale consists of 32 items and 4 subsections. According to the internal consistency method used in the development phase of the "Ostomy Self-Care Index" scale, Cronbach's alpha value was found to be 0.965 for the sub-scales, 0.965 for "Self-Care Maintenance", 0.953 for "Self-Care Monitoring", 0.930 for "Self-Care Management", 0.962 for "Self-Care Confidence" and 0.975 for the total. As a result of the factor analysis, "Self-Care Monitoring" and "Self-Care Confidence" sub-dimensions were grouped under a single factor.
Pittman Ostomy Complication Severity Index | Average 3 months after completion of stoma care education.
  Stoma complications experienced by patients with stoma will be evaluated. The scale was developed by Pittman et al. 2014 to assess the severity of ostomy complications in the postoperative period. The Turkish validity and reliability of the scale was conducted by Aslantaş et al. in 2020. Each item of the Likert-type scale consisting of 9 items is evaluated in the range of 0-3 points. Each item includes one of the stoma complications: leakage, peristomal irritant dermatitis, pain, bleeding, stomal necrosis, stomal stenosis, retraction, mucocutaneous separation and hyperplasia. A score of ''0'' indicates no complications and ''3'' indicates very serious complications. The total score for all items is a minimum of ''0'' and a maximum of ''27''. The highest total score indicates a very serious complication. The scale has no sub-dimensions.
Peristomal Skin Tool | Average 3 months after completion of stoma care education.
  The peristomal skin tool was developed in 2009 with the collaboration of 12 expert stoma care nurses from different countries, dermatologist recommendations and the support of Coloplast A.Ş. (Humlebaek, Denmark). The tool consists of two parts; Color change, Erosion, Uncontrolled tissue growth score calculation guide and Assessment, Intervention, Monitoring guide. The validity and reliability of the tool in our country was conducted by Harputlu and Özsoy in 2016. The intraobserver agreement coefficient of the peristomal skin tool was reported to be very good (0.83-1) and the interobserver agreement coefficient was reported to be moderate to good (0.51-0.77).
Ostomy Adjustment Inventory-23 | Average 3 months after completion of stoma care education.
  It is a 23-item self-assessment scale developed by Simmons et al. to determine the level of stoma adaptation of individuals with stoma. The Turkish validity and reliability of the scale was conducted by Karadağ et al. in 2011. The 23-item self-report scale consists of 4 sub-factors including acceptance (items 1, 3, 4, 6, 9, 14, 15, 19, 23), anxiety/worry (items 12, 13, 17, 20, 21), social adjustment (items 5, 7, 8, 11) and anger (items 2 and 10). In addition, 3 items (16, 18 and 22) were not included in any sub-factor. Each item in the scale is evaluated on a 5-point Likert scale (0-4 points; Strongly agree, Agree, Not sure, Disagree, Strongly disagree) and the higher score obtained from each item indicates an increase in compliance. Twelve items in the scale (items 2, 5, 7, 8, 10, 11, 12, 12, 13, 16, 17, 18 and 21) are reverse scored because they contain negative statements.
Computer System Usability Questionnaire | Average 3 months after completion of stoma care education.
  The scale will be used to determine the ability of patients receiving mobile-based stoma education to use the educational content. "Computer System Usability Questionnaire was developed by Lewis in 1995. The Turkish validity and reliability of the questionnaire was conducted by Erdinç and Lewis in 2013. The questionnaire categorizes the usability of a computer system into the dimensions of system usefulness, information quality and interface quality. The Turkish form is a short version of the questionnaire and consists of 13 items. Each item is scored from 1 (Strongly agree) to 7 (Strongly disagree). Alpha correlation coefficients of the Turkish version of the scale were calculated between 0.73 and 0.92.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University Faculty of Nursing, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ambe PC, Kurz NR, Nitschke C, Odeh SF, Moslein G, Zirngibl H. Intestinal Ostomy. Dtsch Arztebl Int. 2018 Mar 16;115(11):182-187. doi: 10.3238/arztebl.2018.0182. PMID 29607805
- [Background] Azer SA, AlKhawajah NM, Alshamlan YA. Critical evaluation of YouTube videos on colostomy and ileostomy: Can these videos be used as learning resources? Patient Educ Couns. 2022 Feb;105(2):383-389. doi: 10.1016/j.pec.2021.05.023. Epub 2021 May 18. PMID 34045092
- [Background] Azodo, Clement C., and Vivian O. Omuemu. 2017. "Perception of Spirituality, Spiritual Care, and Barriers to the Provision of Spiritual Care among Undergraduate Nurses in the University of Lagos, Nigeria." Journal of Clinical Sciences 14(1):119-25. doi: 10.4103/jcls.jcls.
- [Background] Capilla-Diaz C, Bonill-de Las Nieves C, Hernandez-Zambrano SM, Montoya-Juarez R, Morales-Asencio JM, Perez-Marfil MN, Hueso-Montoro C. Living With an Intestinal Stoma: A Qualitative Systematic Review. Qual Health Res. 2019 Jul;29(9):1255-1265. doi: 10.1177/1049732318820933. Epub 2019 Jan 25. PMID 30678525